CLINICAL TRIAL: NCT06302946
Title: Effect of Neuromuscular Stimulation and Mindfulness Breathing on Pulmonary, Physical Functions and Stress in Patients With Stroke
Brief Title: Effect of Neuromuscular Stimulation and Mindfulness Breathing in Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005024
Record Dates: First submitted 2024-02-14; First posted 2024-03-12 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): will receive neuromuscular stimulation and mindfulness breathing
  Interventions: Other: neuromuscular stimulation and mindfulness breathing
- control group (Active Comparator): The control group will receive neuromuscular stimulation only.
  Interventions: Other: neuromuscular electrical stimulation

INTERVENTIONS:
Other: neuromuscular stimulation and mindfulness breathing — Receive neuromuscular stimulation and mindfulness breathing; the experimental group participants will receive neuromuscular electrical stimulation with Mindful breathing.
  Arms: experimental group
Other: neuromuscular electrical stimulation — participants in the control group perceived neuromuscular electrical stimulation
  Arms: control group

SUMMARY:
It is an interventional study in which 60 stroke patients were estimated to enroll according to random allocation and divided into two groups. The experimental group will receive neuromuscular stimulation and mindfulness breathing, while the control group will receive neuromuscular stimulation only.

DETAILED DESCRIPTION:
It is an interventional study in which 60 stroke patients will be estimated to enroll according to random allocation and divided into two groups. The experimental group will receive neuromuscular stimulation and mindfulness breathing, while the control group will receive neuromuscular stimulation only. The experimental group participants will receive neuromuscular electrical stimulation that will last 12 consecutive weeks, three sessions per week protocol with Mindful breathing is a mindfulness exercise that involves using breathing as an object of attention.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:
* All Patients of this study will be diagnosed as stroke and the diagnosis will be confirmed by computed tomography or MRI (El-Tamawy et al., 2021).
* Age of patients will be ranged from 50 to 65years (males and females).
* All patients will be hemodynamically stable.
* Patients with good cognition that enables them to understand the requirements of the study.

Exclusion Criteria:

* • The potential participants will be excluded if they meet one of the following criteria:

  * Patients who cannot follow instructions as sensory aphasia, blindness, dementia, and deafness.
  * Patients with any orthopedic, neurological, or chest disorders that affect trunk muscles control or cause respiratory disorders as COPD.
  * Patients with cognitive and psychiatric disorders.
  * Patients with unstable cardiovascular conditions.
  * Patients with contraindications to neuro electrical stimulation as:
  * Cardiac pace maker.
  * Acute abdominal surgery.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ventilatory function | 12 weeks
  By a spirometer, forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), the ratio of forced vital capacity to forced expiratory volume (FEV1/FVC), and peak expiratory flow will be measured.

SECONDARY OUTCOMES:
level of stress | 12 weeks
  perceived stress questionnaire Individual scores on the perceived stress questionnaire can range from 0 to 40 with higher scores indicating higher perceived tress
Functional independence measure | 12 weeks
  The Functional independence measure consists of 18 measures organized into six dimensions and ranges from 18 to 126
level of physical function | 12 weeks
  short physical performance battery group of measures that combines the results of the gait speed, chair stand and balance tests

CONTACTS AND LOCATIONS:
Overall Officials: marwa elsayed, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing with other researches
Supporting Information: Study Protocol
Time Frame: 12 months
Access Criteria: after acceptance of publishing journal
URL: https://www.ekb.com